CLINICAL TRIAL: NCT05445674
Title: Plasma Exchange Therapy for Post- COVID-19 Condition: A Pilot, Randomized Double-Blind Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: IrsiCaixa (Other); Banc de Sang i Teixits (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAX
Record Dates: First submitted 2022-06-27; First posted 2022-07-06 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Post-COVID19 Condition
Keywords: SARS-CoV-2; COVID-19; Long COVID19; Plasma exchange (PE); Plasmapheresis
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Plasmapheresis

STUDY DESIGN:
Intervention Model Description: Prospective, randomized (1:1), double-blind, placebo-controlled study
Who Masked: Participant, Investigator
Masking Description: This will be a double blind, placebo-controlled study. Masking of investigational products will ensure that both the investigator and the participant are blinded to the type of exchange procedure. Patients will be unable to distinguish true from sham procedures at the end of the study. Each procedure will take approximately 2 hours to complete. In the sham procedure, the patients will also underwear 6 procedures lasting approximately 2 hours each. Blinding will be maintained throughout the study until after 3-month follow-up assessment of the last patient exchanged
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma Exchange (Experimental): 6 sessions of PE with human serum 5% albumin. Plasma exchange sessions will occur on days 1, 3, 8, 10, 15 and 17
  Interventions: Combination Product: Plasma Exchange Procedure
- Sham Plasma Exchange (Sham Comparator): 6 sessions of sham plasma exchange (one infusion of sterile saline solution 0.9%) on days 1, 3, 8, 10, 15 and 17.
  Interventions: Other: Sham Plasma Exchange Procedure

INTERVENTIONS:
Combination Product: Plasma Exchange Procedure — Plasma exchanges will be performed with 5% albumin as the replacement fluid. The typical schedule prescribed will be an exchange of 1 volemia. Blood will be separated into cells and plasma; the cells will be combined with reconstituted 5% human serum albumin and reinfused into the patient with normal saline
  Other Names: Plasmapheresis
  Arms: Plasma Exchange
Other: Sham Plasma Exchange Procedure — For sham plasma exchange procedures, a sound behind the curtain will be performed imitating the sound of the cell processing platform. In these cases, only one infusion of 200 to 250ml of sterile saline solution 0.9% will be performed during the time stablished for all procedures. Albumin will not be necessary for those patients in the Sham plasma exchange arm
  Arms: Sham Plasma Exchange

SUMMARY:
PAX is a prospective, randomized (1:1), double-blind, placebo-controlled study, that have as a objective to evaluate the safety and tolerability of plasma exchange (PE) in patients with Post Acute Covid-19 Syndrome (PCC) comparing to sham plasma exchange. The participants will be randomized in two arms: (1) 6 sessions of PE (Plasma Exchange) with human serum albumin 5% or (2) 6 sessions with placebo (infusion of of sterile saline solution 0.9%) on days 1, 3, 8, 10, 15 and 17.

DETAILED DESCRIPTION:
Randomized participants will receive plasma exchange (PE) or sham PE (placebo) (6 sessions: V2, V3, V4, V5, V6 and V7) and will continue their follow-up visits(V8d22, V9d45, V10d90). Plasma volumes will be replaced, which will vary depending on sex, height, weight and hematocrit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female individuals 18 years-old or older.
2. Evidence of previous SARS-CoV-2 infection at least 90 days prior to study recruitment, defined by either (a) Nasopharyngeal SARS-CoV-2 nucleic acid test (Polymerase chain reaction [PCR] or Transcription-Mediated Amplification [TMA] (b) validated Nasopharyngeal Lateral Flow Assay rapid antigen test [RAT], or (c) SARSCoV-2 serology before SARS-CoV-2 vaccination.
3. Symptoms of PCC after 90 days of infection and that last for at least 2 months and cannot explained by an alternative diagnosis.
4. Not able to perform all usual duties/ activities due to symptoms, pain, depression or anxiety, defined as grades 3 or 4 in the post-COVID-19 Functional Status (PCFS) scale.
5. Availability of an adequate peripheral venous cannulation.
6. If women of childbearing potential, use of a highly effective method of contraception (abstinence, hormonal contraception, intra-uterine device [IUD], or anatomical sterility in self).
7. Willing to comply with the requirements of the protocol and available for followup for the planned duration of the study.
8. Has understood the information provided and capable of giving informed consent. Exclusion criteria

Exclusion Criteria:

1. SARS-CoV-2 infection diagnosed during the previous 90 days.
2. Last SARS-CoV-2 vaccine dose during the previous 30 days.
3. No significant limitations in the subject's ability to perform all usual duties/activities (i.e., grades 0, 1 or 2 in PCFS scale).
4. Medical conditions for which 250 mL of intravenous fluid is considered dangerous (i.e., decompensated heart failure or renal failure with fluid overload, among others).
5. Pregnant or breastfeeding women.
6. Contraindications for therapeutic PE: Non-availability of an adequate peripheral venous catheter, hemodynamic instability, septicemia, known allergy to fresh frozen plasma or replacement colloid/albumin, known allergy to heparin.
7. Current or planned hospital admission for any cause during the study follow-up.
8. Inability to consent and/or comply with study requirements, in the opinion of the investigator.
9. Currently participating or planning to participate in any other clinical trial until day 90 of follow-up.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of PE in patients with Post-Acute Covid-19 Syndrome (PCC) comparing to sham plasma exchange (placebo) | Within 90 days from the treatment start
  Proportion of adverse events (AEs) through day 90, considering:
  * All AEs
  * Grade 3 and 4 AEs
  * AEs leading to study discontinuation
Proportion of subjects with Grade 0, 1 o 2 functional disability assessed by the functional status scale (PCFS) | From baseline to day 90
  Grade 0, 1 o 2 functional disability assessed by the functional status scale (PCFS), being 0 the better outcome and 4 the worse outcome
Proportion of subjects with Grade 0, 1 o 2 functional disability assessed by the fatigue severity scale (FSS) | From baseline to day 90
  Grade 0, 1 o 2 functional disability assessed by the fatigue severity scale (FSS), being 1 the better outcome and 70 the worse outcome

SECONDARY OUTCOMES:
Assess the ability of PE to improve PCC symptoms | At days 0, 8, 15, 22, 45 and 90
  Can Ruti PCC symptoms scale questionnare by days 0, 8, 15, 22, 45 and 90
Assess the impact of PE on quality of life in subjects with PCC | At day 0, 8, 15, 22, 45 and 90.
  Quality of life questionnaires: EuroQol-5D questionnaire being 5 the better outcome and 15 the worse outcome.
Assess the impact of PE on quality of life in subjects with PCC using MOS-HIV questionnaire | At day 0, 8, 15, 22, 45 and 90.
  Quality of life questionnaires: MOS-HIV questionnaire being 4 the better outcome and 1 the worse outcome.
Assess the impact of PE on neurocognitive symptoms in subjects with PCC using NeuScreen fluency Test | At days 0, 22 and 90
  The neurocognitive evaluation assessed by the NeuScreen fluency test (Seconds)
Assess the impact of PE on neurocognitive symptoms in subjects with PCC using MEF-30 questionnaire | At days 0, 22 and 90
  The neurocognitive evaluation assessed by the MEF-30 questionnaire, with being 0 the better outcome and 120 being the worse outcome.
Assess the impact of PE on neurocognitive symptoms in subjects with PCC using HADs questionnaire | At days 0, 22 and 90
  The neurocognitive evaluation assessed by the HADs questionnaire, with being 0 as the better outcome and 21 being the worse outcome.
Changes in cellular anti-SARS-CoV-2 immunity associated with PE in subjects with PCC by the determination of SARS-CoV-2 specific igG | At day 0, 8, 15, 22, 45 and 90.
  Changes in cellular anti-SARS-CoV-2 immunity associated with PE in subjects with PCC by the determination of SARS-CoV-2 specific igG in plasma (Arbitrary Units, AU)
Changes in cellular anti-SARS-CoV-2 immunity associated with PE in subjects with PCC by the neutralization activity evaluation | At day 0, 8, 15, 22, 45 and 90.
  Changes in cellular anti-SARS-CoV-2 immunity associated with PE in subjects with PCC by the analysis of reciprocal titers of neutralizing antibodies against SARS-CoV-2
Changes in cellular anti-SARS-CoV-2 immunity associated with PE in subjects with PCC by the T-Cell response | At day 0, 8, 15, 22, 45 and 90.
  Changes in cellular anti-SARS-CoV-2 immunity associated with PE in subjects with PCC by the reduction of T-Cell response (%) from plasma samples
Determination of residual SARS-CoV-2 particles (RNA) in plasma from subjects with PCC | At days 0, 8, 15, 22, 45, and 90
  Virological assessment to determine the residual SARS-CoV-2 RNA (copies/mL)
Changes in microbiota associated with PE in subjects with PCC | At day 1, 8, 15, 22, 45 and 90
  Stool assessment to determine the residual SARS-CoV-2 RNA (copies/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Mateu Pruñonosa, PhD, MD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain

REFERENCES:
- [Derived] Espana-Cueto S, Loste C, Llados G, Lopez C, Santos JR, Dulsat G, Garcia A, Carmezim J, Carabia J, Ancochea A, Fernandez-Prendres C, Morales-Indiano C, Quirant B, Martinez-Caceres E, Sanchez A, Parraga IG, Chamorro A, San Jose A, Abad E, Munoz-Moreno JA, Prats A, Fumaz CR, Coll-Fernandez R, Estany C, Torrano P, Puig J, Clotet B, Tebe C, Massanella M, Paredes R, Mateu L. Plasma exchange therapy for the post COVID-19 condition: a phase II, double-blind, placebo-controlled, randomized trial. Nat Commun. 2025 Feb 24;16(1):1929. doi: 10.1038/s41467-025-57198-7. PMID 39994269